CLINICAL TRIAL: NCT00540553
Title: A Randomized, Double-Blind, Placebo Controlled, Dose Escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of GSK971086 After a Single Dose and 7 Days of Repeat Dosing in Healthy Adult Male Volunteers
Brief Title: Study to Test Safety, Tolerability and Blood Levels of GSK971086 After 1 Dose & 7 Days of Dosing in Healthy Adult Males
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: SAR109935
Record Dates: First submitted 2007-10-04; First posted 2007-10-08 (Estimated); Last update posted 2012-03-19 (Estimated); Status verified 2011-02

CONDITIONS: Healthy Subjects; Androgen Deficiency
Keywords: SARM,; FTIH,; pharmacokinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: placebo
Drug: GSK971086
  Other Names: placebo

SUMMARY:
This research study is the first administration of GSK971086 in humans. The purpose of this study is to assess the safety and tolerability of GSK971086, as well as, how much GSK971086 is in your blood after different doses

ELIGIBILITY:
Inclusion Criteria:

* Males between 18 and 50 years of age (inclusive), at the time of signing the informed consent form.
* Healthy, as determined by the Investigator, based on medical evaluations performed during the Screening Period including medical history, physical examination, clinical laboratory tests, and cardiac monitoring.
* Subjects must agree to use an acceptable method of contraception as described in the protocol. These criteria must be followed from the time of the first dose of study drug until completion of the Final Safety and PK Visit in the Follow-up Period.
* Body weight and Body Mass Index (BMI) within the ranges defined in the protocol.
* Subject is able to understand and comply with protocol requirements, instructions, and protocol-stated restrictions, including those listed in the informed consent form.
* Subject has given informed consent to participate in the study as indicated by providing a signed and dated written informed consent form prior to any study procedures.

Exclusion Criteria:

* Subjects with a history of clinically significant endocrine, gastrointestinal, hepatic,cardiovascular, neurological, haematological, immunological, renal, respiratory, or genitourinary abnormalities or diseases.
* Subjects with a history at any time in the past of coronary artery disease, congestive heart failure, angina, myocardial infarction, any cardiac surgery, valvular heart disease, clinically significant arrhythmia, dyspnea, pulmonary edema, stroke, or transient ischemic attack. ECG exclusion criteria as defined in the protocol.
* Subjects with a history of malignancy that is not in complete remission for at least 5 years, 1 year for non-melatonomatous skin carcinoma.
* Subjects with values outside the specified ranges in the protocol for the following Key Clinical Laboratory Tests must be excluded from the study: liver function tests, renal function, electrolytes, metabolic, muscle and haematology.
* Prostate Specific Antigen (PSA) >3.0ng/mL at Screening or subjects with a family history of early onset prostate cancer or multiple members with prostate cancer.
* History of serious psychological disorders such as schizophrenia, uncontrolled bipolar disorder, and suicidal behaviour.
* History of drug or alcohol abuse within 5 years prior to the Screening Period.
* Positive test for illicit drugs or alcohol during Screening assessments. A minimum list of illicit drugs that will be screened for are listed in the protocol.
* History of regular alcohol consumption averaging >14 drinks/week within 12 months prior to the Screening Period.
* A positive test for Human Immunodeficiency Virus (HIV), Hepatitis B surface antigen, or Hepatitis C antibody upon screening, or at any time prior to the Screening Period.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 14 days or 5 half-lives (whichever is longer) prior to the first dose of study drug, however, the use of acetaminophen, ibuprofen, and naproxen will be allowed, as described in the protocol.
* The subject has participated in a clinical trial and has received a drug or a new chemical entity within 30 days or 5 half-lives, or twice the duration of the biological effect of any drug (whichever is longer) prior to the first dose of current study drug.
* History of drug or other allergy that, in the opinion of the Investigator, contraindicates their participation.
* Where participation in study would result in donation of blood in excess of 500mL within a 56 day period.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Consumption of red wine, Seville oranges, grapefruit or grapefruit juice from 7 days prior to the first dose of study drug until check-out from the clinic on the last day of the Treatment Period.
* Unwillingness to adhere to the study Lifestyle Guidelines as described in the protocol.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 126 (Actual)
Dates: Start 2007-08; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Adverse events: | all visits
hematology, clinical chemistry, urinalysis: | Part A Days -2,2,3,14,28 & Part B Days -2,2,5,8,14,21,35
vital signs & 12-lead ECGs: | Part A Days -2-3,7,28 & Part B Days -2-9,14,35

SECONDARY OUTCOMES:
GSK 971086 Plasma blood level: | art A Days 1,2,3,7,14,21,28 & Part B Days 1-9,14,21,28,35
PBone & muscle biomarkers: | Part A Days 1,2,7,14,21,28 & Part B Days 1,3,8,14,21,28,35

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Evansville, Indiana, United States